CLINICAL TRIAL: NCT04236206
Title: Effectiveness of a Mobile Phone Short Message Service on Glycemic Control and Adherence to Treatment for Type 2 Diabetes
Brief Title: Short Message Service for Type 2 Diabetes
Acronym: SMS4T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: High Institute of Public Health, Egypt (Other)
Responsible Party: Principal Investigator, Rehab A. Rayan, PhD Researcher in the Department of Epidemiology, High Institute of Public Health, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RR-SMS4T2D-2020
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Medication adherence; Telemedicine; mhealth; SMS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Quasi-experimental; non-randomized, pre-test, post-test control group design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS Recipients (Experimental): • Mobile phone SMSs will be sent to the intervention group with the aim of improving medication adherence and knowledge about diabetes, its complications, diet and physical activity.
  Interventions: Behavioral: Mobile Phone Short Message Service
- Non-SMS Recipients (No Intervention): Control group with no intervention.

INTERVENTIONS:
Behavioral: Mobile Phone Short Message Service — SMS content will be adopted from the validated Arabic national and international diabetes educational materials (Centers for Disease Control (CDC), 2018; Diabetes Australia, 2004; Diabetes Queensland, 2012; Utah Diabetes Control Program, 2005).
  * The mobile phone SMSs will be pre-tested for clarity on a sample of 10 patients similar to the study population and their comments on the SMSs wording will be used to modify them to ensure acceptance.
  * The SMS will be sent to participants using the internet, open-source software for bulk messages and a local telephone network provider.
  * Patients will be encouraged to send messages/call the researcher for any queries encountered.
  Arms: SMS Recipients

SUMMARY:
Diabetes is a chronic disease where type 1 diabetes (T1D) is due to autoimmune ẞ-cell destruction, usually leading to absolute insulin deficiency, type 2 diabetes (T2D) is due to a progressive loss of ẞ-cell insulin secretion frequently on the background of insulin resistance. A third type-Gestational diabetes mellitus (GDM)-is diagnosed in the second or third trimester of pregnancy and was not clearly overt diabetes prior to gestation (American Diabetes Association. Lifestyle management can enhance diabetes care and it includes diabetes self-management education and support (DSMES), medical nutrition therapy, physical activity, smoking cessation counselling, and psychosocial care. However, health systems cannot control all the factors that influence a person's overall health, as physicians are unable to check regularly what their patients eat or whether they properly adhere to their medications. Pharmacists involved in DSMES can help patients achieve therapeutic and lifestyle goals. This active participation requires that the pharmacist's practice extend beyond the traditional role. Patients and care providers should work together to optimize lifestyle aspects through the entire care process. Telemedicine "healing at a distance" signifies the use of information and communication technology to improve patient outcomes by increasing access to care and medical information. Using mobile and wireless technologies to achieve health objectives (mHealth) can universally transform health services' delivery. Mobile phones can easily reach population since they have exceeded other communication technologies in Low and middle-Income countries (LMICs). The results of the present study will help the policy-makers in the MOHP to understand the importance of creating healthcare systems that meet the needs of patients and providers and develop DSMES strategy with the help of pharmacist educator and using innovative mobile phone technology.

DETAILED DESCRIPTION:
The global prevalence of diabetes among adults aged over 18 years old has increased from 4.7% in 1980 to 8.5% in 2014 (Mathers & Loncar, 2006; WHO, 2018b). The World Health Organization (WHO) estimates that diabetes was the seventh leading cause of death in 2016 (WHO, 2016; WHO, 2018a). Current national statistics show that around 17% of all Egyptian adults have diabetes, and over 60% of diabetics receive no treatment (Eastern Mediterranean Regional Office (EMRO), 2016). According to the WHO, there will be 6,726,000 cases of diabetes in Egypt by 2030 (WHO, 2000).

Almost 45% of patients with T2D cannot achieve adequate glycemic control (HbA1c <7%). Poor medication adherence in T2D is a common public health problem and is associated with poor glycemic control, increased morbidity and mortality, and increased costs of outpatient care, emergency room visits, hospitalization, and managing complications of diabetes (Polonsky & Henry, 2016).

Pharmacists involved in DSMES can help patients achieve therapeutic and lifestyle goals. This active participation requires that the pharmacist's practice extend beyond the traditional role (Shane-McWhorter et al., 2009). Patients and care providers should work together to optimize lifestyle aspects through the entire care process (Abaza & Marschollek, 2017).

In Egypt, the Ministry of Health and Population (MOHP) is partially implementing diabetes education, mostly in outpatient clinics via educational meetings or counselling with physicians/ nurses. Patients often report difficulty sticking to healthy lifestyles. They are also liable to forget or ignore their physician's advice after leaving the clinic. Therefore, they need an educational method that can easily reach them to make knowledgeable patients and save the physician's critical time (Abaza & Marschollek, 2017).

According to the Ministry of Communications and Information Technology (MCIT) in Egypt, up to October 2019, there were 95.25 million mobile subscriptions as opposed to 8.72 million fixed-line subscriptions (Ministry of Communication and Information Technology [MCIT], 2019). Moreover, there were 38.67 million mobile internet users versus 7.17 million Asymmetric Digital Subscriber Line subscriptions in the same month; the mobile internet users could reflect the proportion of smartphone owners in the country (MCIT, 2019). In contrary to mobile internet or smartphone applications, short message service (SMS) can provide a simple way of communication reaching a larger population since almost all types of mobile phones support them (Abaza & Marschollek, 2017).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old and more.
* Diagnosed with T2D up to 15 years according to the American Diabetes Association (ADA) standards (ADA, 2018).
* With poorly controlled diabetes, (pre-intervention HbA1c values of 7% up to 10%).
* Registered in the selected primary health care (PHC) centers and living in Alexandria.
* Currently on oral medication therapy (if purchased from the center pharmacy) and able to afford the cost for 6 months treatment (if purchased from an external pharmacy).
* Has a personal mobile phone.
* Know how to retrieve/read SMS on the mobile phone (Arabic alphabets).
* Available for the study duration.

Exclusion Criteria:

* Patients with clinical conditions that might interfere with the study such as pregnancy, mental illness, poor eyesight, hearing or vocalization, visual, renal or liver impairment, other serious illness or co-morbidities requiring hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | Change from Baseline HbA1c level at 6 months.
  To assess the effect of the intervention on patients with type 2 diabetes in terms of glycemic control (HbA1c level).

SECONDARY OUTCOMES:
Medication Adherence | Change from Baseline Medication Adherence at 6 months.
  To assess the effect of the intervention on patients with type 2 diabetes in terms of adherence to the prescribed hypoglycemic medications using the short form of adherence to refills and medications scale (ARMS-SF).

OTHER OUTCOMES:
Diabetes-related Knowledge | Change from Baseline Diabetes-related Knowledge at 6 months.
  To assess the effect of the intervention on patients with type 2 diabetes in terms of diabetes-related knowledge (the disease symptoms, its complications, tests, importance of medication adherence, diet, physical activity and regular care) using a predesigned structured interviewing questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A Rayan, PharmD, Principal Investigator — High Institute of Public Health, Alexandria University
Locations (1):
- Family Health Centers, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SMS education for the promotion of diabetes self-management in low & middle-income countries: a pilot randomized controlled trial in Egypt. — https://dx.doi.org/10.1186%2Fs12889-017-4973-5
- See also: G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. — https://doi.org/10.3758/BF03193146
- See also: mHealth interventions to counter noncommunicable diseases in developing countries: still an uncertain promise. — https://doi.org/10.1016/j.ccl.2016.08.009
- See also: Effectiveness of mobile phone short message service on diabetes mellitus management; the SMS-DM study. — https://doi.org/10.1016/j.diabres.2011.07.025
- See also: Projections of global mortality and burden of disease from 2002 to 2030. — https://doi.org/10.1371/journal.pmed.0030442
- See also: Use of mHealth systems and tools for non-communicable diseases in low- and middle-income Countries: a systematic review. — https://doi.org/10.1007/s12265-014-9581-5
- See also: Poor medication adherence in type 2 diabetes: recognizing the scope of the problem and its key contributors. — https://doi.org/10.2147/PPA.S106821